CLINICAL TRIAL: NCT03181984
Title: Postmarketing Safety Study of Hemoporfin in Patients With Port Wine Stain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMME-S1612
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain | interventions — hematoporphyrin monomethyl ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemoporfin (Experimental)
  Interventions: Drug: Hemoporfin

INTERVENTIONS:
Drug: Hemoporfin — Hemoporfin mediated photodynamic therapy

SUMMARY:
This study is to provide safety information of hemoporfin during the post-marketing period as required by China Food and Drug Administration (CFDA) regulations in order to identify any potential drug related treatment factors in the Chinese population, such as unknown/unexpected adverse reactions, the incidence of adverse reactions under the routine drug uses.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 14 to 65 years-old；
* Clinically diagnosed of Port-wine Stain;
* Patients receiving hemoporfin based upon the clinical judgment of the investigator;
* Written informed consent signed and agreed to receive periodic follow-up

Exclusion Criteria:

* Allergy to porphyrins and analogues; Photosensitivity; Porphyria; Allergic constitution;
* Scar diathesis;
* Pregnancy or unwilling to adopt reliable contraceptive measures during the month after drug application;
* Be judged not suitable to participate the study by the investigators

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 96 weeks after hemoporfin application

SECONDARY OUTCOMES:
Satisfaction rating of the overall treatment by subjects | 8, 24 and 96 weeks after hemoporfin application
Satisfaction rating of the overall treatment by investigators | 8 weeks after hemoporfin application
Response rate | 8 weeks after hemoporfin application
  proportion of patients achieving at least some improvement (color blanching from the baseline >= 20%)

CONTACTS AND LOCATIONS:
Overall Officials: Xuejun Zhu, Principal Investigator — Peking University First Hospital; Jining Tao, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.
Locations (7):
- China (7):
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Affiliated Hospital of Hebei Medical College of traditional Chinese Medicine, Shijiazhuang, Herbei
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - PLA Army General Hospital, Beijing
  - Shanghai Dermatology Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No